CLINICAL TRIAL: NCT00869973
Title: Aprepitant in the Prevention of Delayed Emesis Induced by Moderately Emetogenic Chemotherapy (Cyclophosphamide Plus Anthracyclines) in Breast Cancer Patients: a Double-blind Randomized Study
Brief Title: Aprepitant in the Prevention of Delayed Emesis Induced by Cyclophosphamide Plus Anthracyclines in Breast Cancer Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: We terminated the study after enrolling 580/900 patients due to a slow accrual
Sponsor: S. Maria Hospital, Terni (Other)
Responsible Party: Principal Investigator, Roila Fausto, Dr, S. Maria Hospital, Terni
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IGAR-02-2009; 2008-001237-95
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2009-10

CONDITIONS: Emesis
Keywords: aprepitant; delayed emesis; cyclophosphamide plus anthracyclines; breast cancer; antiemetic
MeSH Terms: conditions — Vomiting; Breast Neoplasms | interventions — Aprepitant; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Aprepitant
  Interventions: Drug: Aprepitant
- 2 (Active Comparator): dexamethasone
  Interventions: Drug: dexamethasone

INTERVENTIONS:
Drug: Aprepitant — Aprepitant 80 mg orally: 24 hours after chemotherapy on day 2 and then at 8 am on day 3
  Arms: 1
Drug: dexamethasone — dexamethasone 4 mg orally: 24 hours after chemotherapy and at 8 pm on day 2, then at 8 am and 8 pm on day 3
  Arms: 2

SUMMARY:
The aim of the study is to compare efficacy and tolerability of aprepitant versus dexamethasone in the prevention of delayed emesis induced by moderately emetogenic chemotherapy (cyclophosphamide plus anthracyclines) in breast cancer patients.

DETAILED DESCRIPTION:
This is a phase III, double-blind, randomized trial, to evaluated the efficacy and safety of aprepitant for the prevention of delayed emesis in patients with breast cancer submitted for the first time to chemotherapy with cyclophosphamide plus anthracyclines.

The study will be carried out during the first cycle of chemotherapy.

For the prevention of acute emesis, all patients will receive, before chemotherapy:

* dexamethasone 8 mg iv in 15 minutes, 30 minutes before chemotherapy;
* palonosetron 0.25 mg iv bolus, 30 minutes before chemotherapy
* aprepitant 125 mg orally, 60 minutes before chemotherapy

After 24 hours from chemotherapy administration, patients will be randomized to receive:

A) dexamethasone 4 mg orally: 24 hours after chemotherapy and at 8 pm on day 2, then at 8 am and 8 pm on day 3.

B) Aprepitant 80 mg orally: 24 hours after chemotherapy on day 2 and then at 8 am on day 3.

The patients will receive prochlorperazine suppositories as rescue medication, for important nausea and vomiting (> 2 episodes) during days 1-5 after chemotherapy.

The patients will receive a diary, which includes a Visual Analogue Scale (VAS) for nausea and vomiting evaluation. All patients will fill out the diary in which, for 6 consecutive days (days 1-6), patients will report for each day the number of vomiting episodes, the intensity and duration of nausea, any antiemetic rescue medication and any adverse event and its treatment.

In addition, on day 1 before chemotherapy and then on day 6, patients will fill out the FLIE (Functional Living Index-Emesis), a questionnaire concerning the impact of nausea and vomiting on their quality of life.

Primary end point is the percentage of complete responses (no vomiting and no rescue treatment) on days 2-5 after chemotherapy administration

ELIGIBILITY:
Inclusion Criteria:

* patients with breast cancer, receiving for the first time chemotherapy with cyclophosphamide + anthracyclines (FAC, FEC, AC, EC).
* patients over 18 years old and those who signed informed consent
* adequate contraception if premenopausal women

Every other anticancer drug in the first 24 hours will be administered after the end of cyclophosphamide plus anthracycline.

Exclusion Criteria:

* patients already submitted to chemotherapy
* patients receiving any chemotherapy on days 2-4 after treatment
* patients with concomitant severe diseases or with predisposition to emesis such as intestinal obstruction, active peptic ulcer, hypercalcemia and brain metastases
* contraindications to corticosteroids (i.e., active peptic ulcer or previous bleeding from peptic ulcer
* patients submitted to concomitant radiotherapy or submitted to radiotherapy in the 15 days before chemotherapy or planned to receive radiotherapy during the 8 days after chemotherapy
* patients receiving other concomitant antiemetic treatments or submitted to antiemetic treatments in the 24 hours before chemotherapy
* patients with nausea or vomiting in the 24 hours before chemotherapy
* patients receiving concomitant steroids, except when administered at physiologic doses
* patients receiving concomitant benzodiazepines, except when used for nocturnal sedation
* patients with WBC count <3000/mm3 or platelet count <70000/mm3
* patients who are pregnant or breast-feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2009-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Percentage of complete responses (no vomiting and no rescue treatment) on days 2-5 after chemotherapy administration | 6 days

SECONDARY OUTCOMES:
Evaluation of the impact on quality of life of the two antiemetic regimens | 6 days
Evaluation of the prognostic factors of delayed emesis in patients receiving a combination of aprepitant, palonosetron and dexamethasone for the prevention of acute emesis | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Roila, MD, Principal Investigator — Oncology Division, S. Maria Hospital, Terni, Italy
Locations (1):
- Fausto Roila, Terni, Terni, Italy

REFERENCES:
- [Result] Warr DG, Hesketh PJ, Gralla RJ, Muss HB, Herrstedt J, Eisenberg PD, Raftopoulos H, Grunberg SM, Gabriel M, Rodgers A, Bohidar N, Klinger G, Hustad CM, Horgan KJ, Skobieranda F. Efficacy and tolerability of aprepitant for the prevention of chemotherapy-induced nausea and vomiting in patients with breast cancer after moderately emetogenic chemotherapy. J Clin Oncol. 2005 Apr 20;23(12):2822-30. doi: 10.1200/JCO.2005.09.050. PMID 15837996
- [Result] Roila F, Hesketh PJ, Herrstedt J; Antiemetic Subcommitte of the Multinational Association of Supportive Care in Cancer. Prevention of chemotherapy- and radiotherapy-induced emesis: results of the 2004 Perugia International Antiemetic Consensus Conference. Ann Oncol. 2006 Jan;17(1):20-8. doi: 10.1093/annonc/mdj078. Epub 2005 Nov 28. PMID 16314401
- [Result] Eisenberg P, Figueroa-Vadillo J, Zamora R, Charu V, Hajdenberg J, Cartmell A, Macciocchi A, Grunberg S; 99-04 Palonosetron Study Group. Improved prevention of moderately emetogenic chemotherapy-induced nausea and vomiting with palonosetron, a pharmacologically novel 5-HT3 receptor antagonist: results of a phase III, single-dose trial versus dolasetron. Cancer. 2003 Dec 1;98(11):2473-82. doi: 10.1002/cncr.11817. PMID 14635083
- [Result] Gralla R, Lichinitser M, Van Der Vegt S, Sleeboom H, Mezger J, Peschel C, Tonini G, Labianca R, Macciocchi A, Aapro M. Palonosetron improves prevention of chemotherapy-induced nausea and vomiting following moderately emetogenic chemotherapy: results of a double-blind randomized phase III trial comparing single doses of palonosetron with ondansetron. Ann Oncol. 2003 Oct;14(10):1570-7. doi: 10.1093/annonc/mdg417. PMID 14504060
- [Result] Italian Group For Antiemetic Research. Randomized, double-blind, dose-finding study of dexamethasone in preventing acute emesis induced by anthracyclines, carboplatin, or cyclophosphamide: J Clin Oncol. 2004 Feb 15;22(4):725-9. doi: 10.1200/JCO.2004.09.040. PMID 14966097
- [Result] Italian Group for Antiemetic Research. Dexamethasone alone or in combination with ondansetron for the prevention of delayed nausea and vomiting induced by chemotherapy. N Engl J Med. 2000 May 25;342(21):1554-9. doi: 10.1056/NEJM200005253422102. PMID 10824073
- [Derived] Roila F, Ruggeri B, Ballatori E, Del Favero A, Tonato M. Aprepitant versus dexamethasone for preventing chemotherapy-induced delayed emesis in patients with breast cancer: a randomized double-blind study. J Clin Oncol. 2014 Jan 10;32(2):101-6. doi: 10.1200/JCO.2013.51.4547. Epub 2013 Dec 9. PMID 24323030